CLINICAL TRIAL: NCT07153146
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Single and Multiple Ascending Doses of PN-881 in Healthy Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of PN-881 in Healthy Subjects.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Protagonist Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PN-881-01
Record Dates: First submitted 2025-08-22; First posted 2025-09-03 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteer
Keywords: PN-881

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Part 1 & Part 2 is masked; Part 3, Part 4 and Part 5 are open label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- PN-881 Oral Solution Single Ascending Dose (Experimental): PN-881 Oral Solution Single Ascending Dose
  Interventions: Drug: PN-881 Oral Solution
- Placebo Oral Solution Single Ascending Dose (Placebo Comparator): Placebo single ascending doses
  Interventions: Drug: Placebo
- PN-881 Oral Solution Multiple Ascending Dose (Experimental): PN-881 Multiple Ascending Doses
  Interventions: Drug: PN-881 Oral Solution
- Placebo Oral Solution Multiple Ascending Dose (Placebo Comparator): Placebo, multiple ascending doses
  Interventions: Drug: Placebo
- PN-881 Oral Tablet Single Dose (Experimental): PN-881 oral tablet single dose
  Interventions: Drug: PN-881 Oral Tablet
- PN-881 Oral Tablet Multiple Dose (Experimental): PN-881 oral tablet multiple dose
  Interventions: Drug: PN-881 Oral Tablet

INTERVENTIONS:
Drug: PN-881 Oral Solution — PN-881 Oral Solution
  Arms: PN-881 Oral Solution Multiple Ascending Dose; PN-881 Oral Solution Single Ascending Dose
Drug: PN-881 Oral Tablet — PN-881 oral tablet
  Arms: PN-881 Oral Tablet Multiple Dose; PN-881 Oral Tablet Single Dose
Drug: Placebo — Placebo
  Arms: Placebo Oral Solution Multiple Ascending Dose; Placebo Oral Solution Single Ascending Dose

SUMMARY:
The goal of this study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of PN-881 in healthy adult participants.

DETAILED DESCRIPTION:
PN-881 will be administered in oral solution and tablet formulations, with dosing under fasting or fed conditions depending on the study part.

The study consists of five parts:

Part 1 - Single Ascending Dose (SAD): Randomised, double-blind, placebo-controlled Part 2 - Multiple Ascending Dose (MAD): Randomised, double-blind, placebo-controlled Part 3 - Tablet Formulation Comparison: Open-label, crossover design; participants will receive different oral tablet formulations Part 4 - Effect of Food: Open-label, crossover design to assess the effect of food on the pharmacokinetics of PN-881. Participants will receive PN-881 tablet formulations in fasted and fed conditions.

Part 5 - Dosing Frequency Comparison: Open-label, randomized study comparing once-daily and twice-daily dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female participants of non-childbearing potential, aged 18-65 years inclusive
2. Body mass index (BMI) between 18 and 32 kg/m² (inclusive) at screening
3. Willing and able to comply with all study requirements and provide written informed consent
4. Male participants with female partners of childbearing potential must agree to use highly effective contraception during the study and for 90 days after the last dose

Exclusion Criteria:

1. Clinically significant history or presence of cardiovascular, gastrointestinal, hepatic, renal, neurological, psychiatric, or allergic diseases
2. History of neoplastic disease (except adequately treated non-melanoma skin cancer)
3. Positive test for hepatitis B, hepatitis C, or HIV at screening
4. History of substance abuse or recreational IV drug use within the past 2 years
5. Clinically significant infection or fever (>38°C) within 2 weeks prior to screening
6. Use of any prescription/non-prescription drugs or herbal supplements within 7 days or 5 half-lives before dosing (unless approved by investigator)
7. Supine blood pressure or ECG abnormalities outside protocol-defined ranges
8. Use of tobacco/nicotine products exceeding 5 cigarettes/day or 2 chews/day
9. Consumption of >21 alcohol units/week (males) or >14 units/week (females)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) | Predose to 7 days after last dose
  Evaluate the safety and tolerability of PN-881 in comparison to placebo after single and multiple doses in healthy subjects assessed for severity, seriousness, and relation to the investigational product.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of PN-881 | 48 hours following the first dose and the last dose
  Highest measured plasma concentration of PN-881 following oral administration.
Area under the plasma concentration-time curve (AUC) of PN-881 | Predose to 48 hours after the first and last dose.
  AUC calculated from 0 to infinity.
Levels of biomarker in serum | Day 1 Predose up to 48 hours post (last) dose
  Pharmacodynamics (PD) of PN-881 by means of increase in levels of biomarker by PN-881 after single and multiple oral doses.

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
Phase I study